CLINICAL TRIAL: NCT03047109
Title: Ephedrine Versus Phenylephrine Infusion for Prevention of Spinal Hypotension During Cesarean Section: Effect on Maternal Cardiodynamics and Fetal Circulation: Randomized Double-blind Study
Brief Title: Ephedrine and Phenylephrine for Spinal Hypotension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed F. Mostafa, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Phenylephrine Hypotension
Record Dates: First submitted 2017-02-07; First posted 2017-02-08 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Spinal Hypotension
Keywords: Ephedrine; Phenylephrine; Spinal Hypotension; Cesarean Section; Maternal Cardiodynamics
MeSH Terms: interventions — Phenylephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): Patients will receive Phenylephrine 30 µg/minute by syringe pump infusion for 30 minutes.
  Interventions: Drug: Phenylephrine
- Group E (Active Comparator): Patients will receive Ephedrine 3 mg/ minute by syringe pump infusion for 30 minutes.
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Phenylephrine — 30 patients will receive Phenylephrine 30 µg/minute by syringe pump infusion for 30 minutes.
  Arms: Group P
Drug: Ephedrine — 30 patients will receive Ephedrine 3 mg/ minute by syringe pump infusion for 30 minutes.
  Arms: Group E

SUMMARY:
Spinal anesthesia is widely used as the procedure of choice for cesarean delivery. In comparison to epidural anesthesia it is faster, easier to perform, patients are more comfortable, complication rates are lower, and it is more cost effective. Spinal anesthesia is an accepted technique in elective cesarean sections. However, hypotension, resulted from sympathectomy is a common problem, especially in pregnant women.

Spinal block causes peripheral vasodilation and venous pooling, which may result in maternal hypotension. Maternal hypotension after spinal anesthesia for cesarean delivery, without prophylactic measures, has a very high incidence (80%-100%). Even though highly investigated, spinal induced hypotension remains a major concern, and it has been referred to as the "Holy Grail" of obstetric anesthesia. The detrimental effects of the spinal induced hypotension are maternal and fetal. Maternal effects are nausea, vomiting and dizziness. Hypotension results in reduced uterine and intervillous blood flow with potential fetal hypoxia and acidosis.

Treatment and prevention of hypotension has been the subject of much investigation and controversy. Prophylactic measures include: 1) left lateral tilt, 2) fluid preload, 3) vasopressors,4) low dose spinal anesthesia. A 15° left lateral tilt is used routinely during cesarean section, to prevent aorto-caval compression, however it is not sufficient as a sole method. Left uterine displacement is achieved by tilting the operating table or by placing a wedge under the woman's hip. Aorto-caval compression also may increase the spread of spinal anesthesia. Among the non-pharmacological interventions studied to minimize the incidence of hypotension sitting the patient up for up to 7 min after CSE anesthesia for cesarean section reduced intraoperative ephedrine requirement without affecting the success of the spinal anesthetic. In contrast, sitting up for 9 min resulted in the need for rescue epidural anesthesia without additional benefit.

Phenylephrine Treatment of vascular failure in shock, shock-like states, drug-induced hypotension or hypersensitivity; correction of paroxysmal supraventricular tachycardia; prolongation of spinal anesthesia; vasoconstriction in regional analgesia; maintenance of adequate level of BP during spinal and inhalation anesthesia. It has a number of important attributes for treating spinal hypotension: (i) as an alpha-adrenergic agonist, its mechanism of action directly addresses the decrease in systemic vascular resistance following spinal anesthesia;(ii) phenylephrine has a faster onset of action compared with ephedrine; (iii) ephedrine is associated with a ﬁve-fold increased risk of fetal acidosis; and (iv) ephedrine is more likely to cross the placenta and increase concentrations of lactate, glucose, and catecholamines in the fetal circulation compared with phenylephrine. However, phenylephrine used alone may be accompanied by maternal bradycardia and does not beneﬁt from widespread clinical experience, as does ephedrine do. Thus, phenylephrine has not yet become popular, particularly for prophylactic use. Clinical experience suggests that phenylephrine may be useful in addition to ephedrine when the latter fails to correct hypotension.

Ephedrine sulphate is a potent sympathomimetic that stimulates both α and β receptors and has clinical uses related to both actions. Its peripheral actions, which it owes in part to the release of norepinephrine, simulate responses that are obtained when adrenergic nerves are stimulated. These include an increase in blood pressure, stimulation of heart muscle, constriction of arterioles.

DETAILED DESCRIPTION:
Study design:

A prospective randomized clinical double-blind study using a computer generated randomization will be conducted in a Women's Health Hospital, Assuit University. Neither the doctor "investigator" nor the participant "parturient" will be aware of the group allocation or the drug used. The study drugs will be prepared by one of the supervisor anesthetist (not included in the procedure, observation or in data collection). The study will be carried on 60 parturient scheduled for elective cesarean section under spinal anesthesia. They will be randomly allocated into two equal groups of 30 parturient each:

P group: Phenylephrine 30 µg/minute by syringe pump infusion for30 min. E group: Ephedrine 3 mg/ minute by syringe pump infusion for30 min. The study solutions (vasopressors) will be prepared by another supervisor anesthetist and will be diluted with normal saline (Na Cl 0.9%) to the same total 50 ml volume in a syringe pump.

Pre-intervention Assessment:

All parturient will undergo full pre-anesthetic checkup (according to ASA guidelines) including detailed history, physical and systemic examinations. They will be kept NOP (nil per mouth) 6-8 hours for solids and 2 hours for water and clear fluids.

Parturient in the holding area:

Baseline monitoring readings of the maternal vital signs including HR, NIBP, SpO2 and RR.

Non-invasive Cardiac Output Monitoring:

The patients will positioned in the supine position, with uterine displacement to the left lateral for several minutes and the electrodes of the noninvasive cardiac output monitor are placed to measure cardiac output. Baseline reading of cardiac output will be recorded before any intervention using NCCOM3 cardiodynamic monitor. . From this apparatus we will get HR, EF, CO /CI, SVR

Uterine blood flow evaluation:

Baseline uterine blood flow will be recorded in the holding area and before any intervention using SONO Ace R5 by the obstetric supervisor. Colour Doppler ultrasound will be used to demonstrate the main ascending branches of left and right uterine arteries as they cross over the hypogastric vessels just before they enter the uterus at the uterine-cervical junction. The high pass filter was set at 125 Hz and the uterine artery will be obtained immediately after the crossing of the hypogastric artery. The sample vol¬ume will be placed on the artery with an angle of about 0°. After detection of blood flow and visu¬alization of the waveform of the uterine artery, five blood flow indices will be automatically cal¬culated:

The pulsatility index (PI) (PI=PSV-EDV/TAMXV); The resistance index (RI) (RI=PSV-EDV/PSV); The peak systolic velocity (PSV, units of cm/s); The end-diastolic velocity (EDV, units of cm/s). TAMXV: Time averaged maximum velocity PSV: Peak systolic velocity. EDV: End-diastolic velocity At least three consecutive correctly imaged blood flow velocity waveforms will be analyzed; both right and left uterine arteries diameters will be measured on a perpendicular B-mode view of the longitudinal vessel section at maxi¬mum magnification. Mean values of bilateral uterine RI and PI will be used for statistical analysis.

Then intravenous cannula 18 G will be inserted into forearm vein under local anesthesia and no premeditated drugs will be given to all women. Ringer's Lactate solution 10ml/kg will be infused for all women participating in the study over 20-30-minutes, and then will be transferred to the operating room.

Parturient in the operating room:

The previous monitoring data will be recorded again for the second time (including vital data, maternal non-invasive cardiac output and uterine blood flow). Then the study solutions will be started to infuse according to the previous description ( to prevent hypotension mostly occur with spinal anesthesia during cesarean section).Then subarachnoid block will be carried out under complete aseptic condition while the in the sitting position and the table in the horizontal level using 25 G pencil point spinal needle, intrathecal block will be performed at level of L 3-4 or L 4-5 vertebral interspaces, 12.5 mg (2.5 ml) of hyperbaric bupivacaine 0.5% and 300 ug morphine sulphate will be injected intrathecally at the rate of 1ml/15 second (12) in all parturients for anesthesia. Immediately after end of injection of drugs intrathecally, the parturient will be placed in the supine position with left uterine displacement. Sensory block will be assessed using loss of sensation in response to cold sensation using piece of ice along midclavicular line bilaterally every 2 minutes until reach the level of T5 dermatome.

A third monitoring reading of the vital data, maternal non-invasive cardiac output and uterine blood flow will be taken 15 minutes after spinal block and before the surgical operation (cesarean section) starts.

Intra-operative Assessment:

After subarachnoid block all will be monitored for HR, NIBP, SpO2 and RR every 5 minutes till the end of the surgery. All parturients will be continuously monitored intra-operatively for any episodes of hypotension, hypertension, bradycardia or tachycardia. Hypotension: defined as more than 20% decrease in maternal systolic blood pressure from the baseline. It will be treated with intravenous crystalloid fluid bolus or drug boluses (1 ml) of the study drug according the groupwhen needed. The total dose of drug boluses will be calculated when used. Hypertension defined as more than 29% increase in maternal systolic blood pressure from the baseline, if occurred, drug infusion will be stopped until the effect ends, then the infusion will be started again. If relapse occur for 2 times, the drug infusion will be stopped and the case will be excluded from the study.

Neonatal Evaluation:

Arterial blood sample will be collected from the fetal umbilical cord immediately through double clamp segment after birth (about 10 cm of umbilical cord during clamping will be sufficient to withdraw the sample). Analysis of the fetal umbilical arterial blood gas will be performed. An umbilical blood PH of less than 7.2 will be considered fetal acidosis (19). To assess the acid-base status and oxygenation of the fetus at delivery. Blood is drawn separately with heparinized syringes from both an umbilical artery and umbilical vein from a doubly clamped segment of the umbilical cord. If both umbilical vein and artery blood show low PO2 (below 30 and 15 mmHg) and high pco2 (above 40 and 50 mmHg) , respectively uteroplacental insufficiency was present.

All newborns will be evaluated by pediatrician regarding the APGAR score at 1st. and 5th .minutes of birth.

Study outcomes Primary outcome

1- The difference in maternal cardiac output between the study groups Secondary outcomes

1. The difference in uterine blood flow indices by Doppler
2. The difference of intraoperative maternal vital singes.
3. The rate of occurrence of neonatal morbidity.
4. Complications or side effects of medications.
5. Parturient satisfaction.

Statistical analysis:

Data will be collected and will be analyzed using SPSS version 20 (SPSS, Inc., Chicago, Illinios, USA). Normally distributed numerical data will be presented as mean +_SD, rang, number and percentage. Numerical variables will be compared among the three groups using the Kruskal-Wallis test and Mann-Whitney test. Categorical variables will be compared among the three groups using the Chi-Square test and Fisher's exact test. P-value of less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-35 years.
* ASA physical I-II
* Singleton term pregnancy.
* Elective cesarean section.

Exclusion Criteria:

* Parturient refusal.
* Women with history of cardiac, respiratory, renal, neurologic or endocrine diseases.
* Women with known allergy to amide local anesthetics or any medications used in the study.
* Any contraindications to regional anesthesia e.g. coagulopathy.
* Pre-eclampsia.
* Fetal abnormalities.
* Emergency surgeries.
* Failed or unsatisfactory spinal block.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Maternal Cardiac Output | 30 minutes
  maternal cardiac output will be done using non-invasive thoracic bio-impedance monitor
Uterine Blood Flow | 30 minutes
  uterine blood flow indices will be done using Doppler

SECONDARY OUTCOMES:
APGAR score | 5 minutes
  All newborns were evaluated by a pediatrician regarding the APGAR score at the 1st and 5th minutes after birth.
Complications | 2 hours
  Percentage of patients with any complications will be recorded and treated

CONTACTS AND LOCATIONS:
Overall Officials: HAMDY A. YOUSSEF, MD, Study Chair — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided